CLINICAL TRIAL: NCT02757820
Title: A Randomized Comparison of Pediatric I-gel, Air-Q With Classic Laryngeal Mask Airway in Terms of Clinical Performance and Fiber Optic Glottic View
Brief Title: A Randomized Comparison of Pediatric I-gel, Air-Q With Classic Laryngeal Mask Airway
Acronym: I-gelvsAir-q
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/ref. 89
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia
Keywords: anesthesia; airway; laryngeal mask airway; I-gel; Air-Q

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LMA classic (Active Comparator): Patients will be anesthetized using Classic laryngeal mask airway that will be inserted lubricated with partially deflated cuff. After insertion, the cuff will be inflated with the recommended volume of air.
  Interventions: Device: LMA Classic
- I-gel (Active Comparator): Patients will be anesthetized using I-gel LMA with its lubricated cuff inserted along the hard palate until resistance is felt, as recommended by the manufacturer.
  Interventions: Device: i- gel
- Air-Q (Active Comparator): Patients will be anesthetized using Air-Q_ ILA, with its lubricated cuff inserted along the hard palate until resistance is felt, as recommended by the manufacturer.
  Interventions: Device: Air-Q

INTERVENTIONS:
Device: LMA Classic — Patients will be anesthetized using Classic laryngeal mask airway that will be inserted lubricated with partially deflated cuff. After insertion, the cuff will be inflated with the recommended volume of air.
  Arms: LMA classic
Device: i- gel — Patients will be anesthetized using I-gel LMA with its lubricated cuff inserted along the hard palate until resistance is felt, as recommended by the manufacturer.
  Arms: I-gel
Device: Air-Q — Patients will be anesthetized using Air-Q_ ILA, with its lubricated cuff inserted along the hard palate until resistance is felt, as recommended by the manufacturer.
  Arms: Air-Q

SUMMARY:
The aim of this randomized trial will be to evaluate the clinical performance of the I-gel, air- Q ILA compared with the LMA classic in pediatric patients undergoing peripheral surgery under general anesthesia.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) Classic has gained popularity for airway management in both anesthesia and resuscitation due to its ease of use. However, insertion of the LMA Classic is not always easy in children due to differences in airway anatomy compared with adults, and more complications are related to its use in younger children compared with adults.

The i-gel has been commercially available in sizes suitable for children since 2010. It has a non-inflatable cuff and an additional lumen for the active or passive drainage of gastric contents (except in size 1). It is available in four children's sizes (1, 1.5, 2 and 2.5).

The air-Q_ ILA, is easily inserted with the index finger of the right hand, while the anesthetist performed jaw's lift with left hand, without a rotational technique (Jagannathan N et al., 2011, Dar long et al, 2014 and Keil et al, 2015).

Oropharyngeal leak pressure is defined as the airway pressure at which air leaks into the mouth or enters the stomach (Hughes et al., 2012). This feature is the most common primary outcome parameter used to evaluate the safety and efficacy of supraglottic airway devices because high pressures generally indicate that adequate ventilation can be achieved without air leakage during positive pressure ventilation at high inspiratory pressures (Teoh et al., 2010).

ELIGIBILITY:
Inclusion Criteria:

Weight: 15-30 kg. Age: 2-9 years. Sex: both males and females. ASA physical status: 1-3. Operation: elective outpatient surgery in which airway management with a LMA would be appropriate.

Exclusion Criteria:

Active respiratory illness (cough, fever, rhinorrhea) on the day of anesthesia, Potentially difficult airway. Patients with history of neck, respiratory, or digestive tract pathology. Patients with gastroesophageal reflux, gastrointestinal stenosis or stricture

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Airway leak pressure | intraoperative
  Airway leak pressure will be determined by closing the adjustable expiratory pressure-limiting (APL) valve and setting the fresh gas flow rate to 3 L/min. The airway pressure at which an audible leak in the mouth is heard is recorded as the "leak pressure". If leak pressure reached 35 cmH2O, the expiratory valve will be opened. After adjusting the APL valve to 35 cmH2O, the maximum tidal volume (TVmax) will be measured by squeezing the balloon of anesthesia circuit until an audible leak occurred. Airway pressures were not allowed to exceed 35 cmH2O.

SECONDARY OUTCOMES:
Fiberoptic laryngoscopic view | intraoperative
  Fiberoptic images will be recorded using a digital camera and will be stored on a personal computer for grading by an independent anesthetist. The images will be graded with a score from 1 to 5, which has been defined and proposed previously (Beringer et al, 2011 and Lee et al, 2012); (grade 1-only larynx seen; grade 2-larynx and epiglottis posterior surface seen; grade 3-larynx and epiglottis tip of anterior surface seen, <50%visual obstruction of epiglottis to larynx; grade 4-epiglottis down folded and its anterior surface seen, >50%visual obstruction of epiglottis to larynx; and grade 5-epiglottis down folded and larynx cannot be seen directly).
ventilation score | intraoperative
  the ventilation score which is scored from 0 to 3 based on three criteria: no leakage with an airway pressure of 15 cm H2O, bilateral chest excursions with a peak inspiratory pressure of 20 cm of H2O, and a square wave capnogram, with each item scoring 0 or 1 point (Sanuki et al., 2011). Thus, if all three criteria are satisfied, the ventilation score is 3.
Heart rate | intraoperative
  the heart rate will be recorded from the monitor screen noninvasively.
peripheral arterial oxygenation | intraoperative
  the peripheral arterial oxygenation will be recorded non invasively from pulse oximeter placed in the finger

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assistant professor, anesthesia department, faculty of medicine, Assiut university
Locations (1):
- Assiut university Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided